CLINICAL TRIAL: NCT00563810
Title: An Ascending Multiple Dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of MYO-029 Administered Intravenously as a 30-Minute Infusion to Healthy Subjects
Brief Title: Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of MYO-029
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 3147K1-103
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Healthy
Keywords: Adult; Aged
MeSH Terms: interventions — Stamulumab

INTERVENTIONS:
Drug: MYO-029

SUMMARY:
This is a multiple dose study assessing the safety, tolerability, pharmacokinetics and pharmacodynamics of an investigational new drug.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 45 years inclusive on study day 1.
* Elderly men and women aged 65 to 80 years inclusive on study day 1.
* Women must be postmenopausal for > or = 1 year (with estradiol < 25 pg/mL and an FSH > 40 mIU/mL).
* Healthy as determined by the investigator on the basis of medical history, physical examination, vital signs, clinical laboratory test results, and 12-leave electrocardiogram.
* Elderly subjects may have stable, nonclinically significant abnormalities on physical examination, and laboratory evaluation.
* Non-smoker.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2004-10; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer